CLINICAL TRIAL: NCT01586793
Title: A Randomized Trial Comparing the Effectiveness and Tolerability of High and Low Frequency Repetitive Transcranial Magnetic Stimulation for Treating Resistant Bipolar Depression: An Exploratory Study
Brief Title: Repetitive Transcranial Magnetic Stimulation for Treating Resistant Bipolar Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, MARCELO T. BERLIM, Director, Neuromodulation Research Clinic, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rTMS-ERB12/05-2012
Record Dates: First submitted 2012-04-24; First posted 2012-04-27 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Bipolar Depression
Keywords: Repetitive transcranial magnetic stimulation; Bipolar depression; Randomized trial; rTMS; Neuromodulation
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Frequency rTMS (Experimental): 10 Hz in 75 trains of 4-seconds duration, with 26-seconds intertrain intervals (3,000 pulses per session) at 120% of the rMT.
  Interventions: Device: Magstim Rapid2 Stimulator
- Low Frequency rTMS (Experimental): 1 Hz in 1 train of 20-minute duration (1,200 pulses per session) at 120% of the rMT.
  Interventions: Device: Magstim Rapid2 Stimulator

INTERVENTIONS:
Device: Magstim Rapid2 Stimulator — 1 Hz in 1 train of 20-minute duration (1,200 pulses per session) at 120% of the rMT.
  Other Names: 1 Hz rTMS
  Arms: Low Frequency rTMS
Device: Magstim Rapid2 Stimulator — 10 Hz in 75 trains of 4-seconds duration, with 26-seconds intertrain intervals (3,000 pulses per session) at 120% of the rMT.
  Other Names: 10 Hz rTMS
  Arms: High Frequency rTMS

SUMMARY:
The aim of this randomized, single-blind trial is to evaluate the effectiveness and tolerability of high frequency or low frequency repetitive transcranial magnetic stimulation (rTMS) in patients with resistant bipolar depression. Patients will be assigned to receive either high or low frequency rTMS for 20 consecutive workdays (4 weeks). 10 Hz (high) frequency rTMS and 1 Hz (low) frequency rTMS will be given over the left or right dorsolateral prefrontal cortex (DLPFC), respectively. Patients will be assessed with several psychometric instruments at baseline, and at weeks 5 and 9.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 70 years
* Current major depressive episode (MDE) in the context of a bipolar disorder type I or II (according to the DSM-IV-TR) that has not improved after more than 2 adequate pharmacological trial(s) in the current episode (failure is defined as a lack of significant clinical improvement after the use of standard mood stabilizers, atypical antipsychotics and/or antidepressants given at their minimum effective dosage or higher for at least 4 weeks of duration)
* Baseline score ≥ 13 on the Quick Inventory of Depressive Symptomatology - Clinician-Administered (QIDS-C), i.e., a MDE of at least moderate intensity

Exclusion Criteria:

* Psychotic features in the current episode
* Lifetime history of a non-mood-related psychotic disorder
* Substance or alcohol abuse/dependence in the past 6 months
* Unstable medical disease (e.g., cardiovascular, renal)
* Presence of mood cycles of < 30 days duration
* Pregnancy and/or lactation
* Presence of a specific contraindication for rTMS (e.g., personal history of epilepsy or convulsion, metallic head implant)
* Hearing loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Week 5
  Pre-post neuromodulation treatment reduction on the scores of the MADRS

SECONDARY OUTCOMES:
21-item Hamilton Depression Rating Scale (HAM-D21) | Week 5
  Response to treatment will be defined as a higher than 50% reduction in pretreatment symptoms severity as measured by the mean HAM-D21 score. Remission will be considered as a HAM-D21 score ≤ 8.
Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) | Week 5
  Response to treatment will be defined as a higher than 50% reduction in pretreatment symptoms severity as measured by the mean QIDS-SR score. Remission will be considered as a QIDS-SR score ≤ 5.
Quick Inventory of Depressive Symptomatology - Clinician (QIDS-C) | Week 5
  Response to treatment will be defined as a higher than 50% reduction in pretreatment symptoms severity as measured by the mean QIDS-C score. Remission will be considered as a QIDS-C score ≤ 5.
Montogmery-Asberg Depression Rating Scale (MADRS) | Week 5
  Response to treatment will be defined as a higher than 50% reduction in pretreatment symptoms severity as measured by the mean MADRS score. Remission will be defined as a MADRS score ≤ 6.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Berlim, MD, MSc, Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Neuromodulation Research Clinic, Douglas Mental Health University Institute, Verdun, Quebec, Canada

REFERENCES:
- [Background] Dell'Osso B, Mundo E, D'Urso N, Pozzoli S, Buoli M, Ciabatti M, Rosanova M, Massimini M, Bellina V, Mariotti M, Altamura AC. Augmentative repetitive navigated transcranial magnetic stimulation (rTMS) in drug-resistant bipolar depression. Bipolar Disord. 2009 Feb;11(1):76-81. doi: 10.1111/j.1399-5618.2008.00651.x. PMID 19133969
- [Background] Dolberg OT, Dannon PN, Schreiber S, Grunhaus L. Transcranial magnetic stimulation in patients with bipolar depression: a double blind, controlled study. Bipolar Disord. 2002;4 Suppl 1:94-5. doi: 10.1034/j.1399-5618.4.s1.41.x. No abstract available. PMID 12479689
- [Background] Nahas Z, Kozel FA, Li X, Anderson B, George MS. Left prefrontal transcranial magnetic stimulation (TMS) treatment of depression in bipolar affective disorder: a pilot study of acute safety and efficacy. Bipolar Disord. 2003 Feb;5(1):40-7. doi: 10.1034/j.1399-5618.2003.00011.x. PMID 12656937